CLINICAL TRIAL: NCT04994470
Title: Evaluation of a Web-based Self-help Intervention Based on Principals of Positive Psychology for Adolescents With Acute or Remitted Major Depressive Disorder
Brief Title: Web-based Self-help Intervention for Adolescents With Acute or Remitted Major Depressive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: Prof. Otto Beisheim Foundation (Other)
Responsible Party: Principal Investigator, Ellen Greimel, Postdoctoral Researcher, Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20114
Record Dates: First submitted 2021-07-30; First posted 2021-08-06 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Depression; Depressive Disorder; Depressive Symptoms; Depressive Disorder, Major
Keywords: Depression; Adolescence; Youth; Web-based Intervention; Self-help; Positive Psychology; Depressive Symptoms; Treatment; Positive Thinking
MeSH Terms: conditions — Depression; Depressive Disorder; Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: Participants are assigned to two groups in parallel for the duration of the study
Who Masked: Participant
Masking Description: Participants are not aware of the assigned intervention group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Web-based intervention group (Experimental): Two-week web-based intervention
  Interventions: Behavioral: Two-week web-based self-help intervention based on principles of positive psychology
- Web-based control group (Sham Comparator): Two-week web-based sham comparator
  Interventions: Behavioral: Two-week web-based text messages containing fun facts

INTERVENTIONS:
Behavioral: Two-week web-based self-help intervention based on principles of positive psychology — The web-based self-help intervention consists of 14 exercises based on the following positive psychology domains: personal strengths, pleasure, gratitude, engagement (flow, mindfulness) and positive relationships.
  The (partly interactive) exercises are created to be implemented by the participants themselves without support of a therapist.
  Before starting the intervention, the participants are told that they will receive a daily email with an instruction for a short exercise over the period of two weeks. The participants are instructed to complete the exercises every day and are told that they will be asked to evaluate these exercises at the next appointment (post-test, week 2).
  Arms: Web-based intervention group
Behavioral: Two-week web-based text messages containing fun facts — The web-based sham comparator consists of 14 text messages containing random interesting facts ("fun facts").
  Before starting the sham comparator, the participants are told that they will receive a daily email with a text message to read every over the period of two weeks. The participants are instructed to read these text messages every day and are told that they will be asked to evaluate these exercises at the next appointment (post-test, week 2).
  Arms: Web-based control group

SUMMARY:
This study aims to evaluate the feasibility and effectiveness of a web-based self-help intervention in adolescents with acute or remitted major depressive disorder. We will examine whether this intervention improves positive affect, reduces stress and alleviates negative affect and depressive symptoms in adolescents aged 12 to 18 years. We will also investigate the rates of adherence among the adolescents who use this web-based intervention and the acceptability of the intervention with adolescents.

DETAILED DESCRIPTION:
Youth with major depressive disorder often have little knowledge about depression, and do not receive an appropriate treatment. Besides little knowledge, concerns about social stigma, confidentiality and limited access to mental health services are some of the main barriers to seek help. Therefore, highly acceptable and easily accessible information and services as a complementary strategy to mental health treatment, such as knowledge about depression and self-help strategies, are urgently needed for young people seeking help for depression.

We developed a website, which provides evidence-based information about depression (e.g., identification, etiology, treatment, and prevention of depression) and will be launched in autumn 2021. Furthermore, the website provides information about self-help strategies (e.g., reducing stress, doing exercise, undertaking positive activities), which are meant to serve as an addition to professional treatments of depression or to promote mental health in adolescents. Target groups of the website are adolescents aged 12 to 18 years seeking help for depression, as well as healthy adolescents seeking information about mental health promotion or depression.

To increase the acceptability of the website and the engagement of young people, the website will integrate continuously updating content consisting of short exercises based on principles of positive psychology. This web-based self-help intervention is thought to provide a mode of delivery (the combination: "online" & "positive psychology"), which is acceptable and engaging to youth. In addition, the provided self-help exercises might be a complementary approach to professional treatments of depression.

Since the website targets two different groups, we will evaluate the web-based self-help intervention accordingly:

Target group 1: Adolescents with a major depressive disorder (acute or remitted) Target group 2: Healthy Adolescents (no mental health condition)

The current study will focus on target group 1. A study focusing on target group 2 can be found in a separately registered clinical trial on clinicaltrials.gov.

The primary aim of the study is to evaluate the feasibility and effectiveness of this web-based self-help intervention to improve positive affect, reduce stress and alleviate negative affect and depressive symptoms in adolescents with acute or remitted depressive disorder.

Participating young people will be randomized to either the web-based intervention group or the web-based control group (i.e. sham intervention / comparator). All participants will be evaluated at pre- and post-intervention, and at a two-week follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Current or remitted diagnosis of MD (ICD-10 diagnoses F32.0; F32.1; F32.2, F33.0, F33.1, F.33.2)
* Intelligence quotient (IQ) of ≥ 80

Exclusion Criteria:

* Acute suicidality
* Schizophrenic disorder
* Pervasive developmental disorder
* Bipolar disorder
* Borderline personality disorder
* Substance dependence disorder
* Insufficient knowledge of German

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 86 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2022-05-02 (Actual); Study Completion 2022-05-02 (Actual)

PRIMARY OUTCOMES:
Beck Depression Inventory - Second Edition (BDI-II) | Pre-test (week 0), post-test (week 2), follow-up (week 4)
  The BDI-II is a self-report inventory to assess the severity of depressive symptoms, rated on a 4-point response scale, with higher scores indicating more severe depressive symptoms. Participants will complete the BDI-II at pre-, post-test and follow-up to determine change in depressive symptoms
Positive and Negative Affect Schedule for Children-Short Form (PANAS-C-SF) | Pre-test (week 0), post-test (week 2), follow-up (week 4)
  The PANAS is a self-report inventory to assess positive and negative affect (10 items for PA and 10 items for NA), rated on a 5-point response scale, with higher scores indicating more positive affect or negative affect. Participants will complete the PANAS at pre-, post-test and follow-up to determine change in negative and positive affect
Perceived Stress Scale (PSS-10) | Pre-test (week 0), post-test (week 2), follow-up (week 4)
  The PSS-10 is a self-report inventory to assess perceived stress, rated on a 5-point response scale, with higher scores indicating more perceived stress. Participants will complete the PSS-10 at pre-, post-test and follow-up to determine change in perceived stress.

SECONDARY OUTCOMES:
Adherence | Post-test (week 2)
  A self-report inventory, designed by the investigators, to measure the rate of adherence to the intervention
Acceptance | Post-test (week 2)
  : A self-report inventory, designed by the investigators, to measure the acceptability / appeal of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Gerd Schulte-Körne, Professor, Study Director — Department of Child and Adolescent Psychiatry, Psychosomatics and Psychotherapy, University Hospital Munich
Locations (1):
- Department of Child and Adolescent Psychiatry, Psychosomatics and Psychotherapy, University Hospital Munich, Munich, Germany, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No
Data in our study contains sensitive patient information, such as sociodemographic information and comorbidities. Since patients could possibly be identified by making our raw data publicly available, ethical principles of protecting patient confidentiality would be breached. Aggregated group data can be made available upon request.